CLINICAL TRIAL: NCT00964171
Title: A Phase II Trial to Assess the Efficacy of Efavirenz as Second-line Monotherapy for the Treatment of Advanced Pancreatic Adenocarcinomas.
Brief Title: Efavirenz as Second-Line Therapy in Treating Patients With Metastatic Pancreatic Cancer
Acronym: PANTER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000641759; IB-PANTER; IB 2008-33; INCA-RECF0888; EUDRACT-2008-004273-18
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — efavirenz

ARMS (1):
- Efavirenz (Other): Efavirenz will be provided by the sponsor as follows: capsule of efavirenz 200 mg. A bottle contains 90 capsules. Investigator will dispense efavirenz to the patients according to the dose adjustment. Each patient will receive efavirenz 600 mg/day until morphological progression. Study drug will be taken every day by oral route at bedtime and in fast condition (1-2 hours far from dinner).
  Interventions: Drug: Efavirenz 600mg

INTERVENTIONS:
Drug: Efavirenz 600mg

SUMMARY:
RATIONALE: Efavirenz may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well efavirenz works as second-line therapy in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy of efavirenz as second-line monotherapy, in terms of non-morphological progression at 2 months, in patients with metastatic adenocarcinoma of the pancreas.

Secondary

* Evaluate non-morphological progression in these patients at 4 months.
* Evaluate non-biological progression in these patients at 2 and 4 months.
* Evaluate the quality of life of these patients at 2 and 4 months.
* Evaluate the overall, progression-free, and event-free survival of these patients.
* Evaluate the tolerability and safety profile of efavirenz in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral efavirenz once daily in the absence of disease progression or unacceptable toxicity.

Patients complete quality-of-life questionnaires using the QLQ-C30 at baseline and at 2 and 4 months.

After completion of study therapy patients are followed up every 2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas

  * No other histological types
* Radiologically confirmed metastatic disease in a non-irradiated area
* Measurable disease according to RECIST criteria
* Must have exhausted first-line gemcitabine hydrochloride chemotherapy
* No CNS metastases

PATIENT CHARACTERISTICS:

* WHO performance status (PS) 0-2 OR Karnofsky PS 70-100%
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Creatinine ≤ 1.25 times upper limit of normal
* Alkaline phosphatase < 5 times normal
* Bilirubin < 3 times normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Has French Social Security in compliance with the French law relating to biomedical research
* Able to comply with study treatment and follow-up
* No severe renal failure
* No severe hepatic impairment
* No known hypersensitivity to the study drug and its excipients
* No depression with a total score of ≥ 13 on the Hospital Anxiety and Depression (HAD) scale
* No active diarrhea that may affect the ability to absorb the study drug
* No other cancer within the past 5 years except carcinoma in situ of the cervix or basal cell carcinoma of the skin
* No geographical, psychiatric, social, or psychological reason that would preclude compliance with study procedures

PRIOR CONCURRENT THERAPY:

* Recovered from all prior anticancer therapy
* More than 30 days since prior investigational drugs and/or participation in a clinical trial
* Prior adjuvant chemotherapy (one-line only) and/or radiotherapy allowed
* No prior enrollment on this study
* No prior treatment acting on the signal transduction pathway
* No prior yellow fever vaccine
* No other concurrent second-line therapy
* No concurrent terfenadine, astemizole, cisapride, midazolam, triazolam, pimozide, bepridil, rye alkaloids, voriconazole, or St. John wort (Hypericum perforatum)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Fonck, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Efavirenz: Efavirenz will be provided by the sponsor as follows: capsule of efavirenz 200 mg. A bottle contains 90 capsules. Investigator will dispense efavirenz to the patients according to the dose adjustment. Each patient will receive efavirenz 600 mg/day until morphological progression. Study drug will be taken every day by oral route at bedtime and in fast condition (1-2 hours far from dinner).
  Efavirenz 600mg
Period: Overall Study
Arm/Group | Efavirenz
Started | 19
Completed | 14
Not Completed | 5
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Arm/Group | Efavirenz
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 56 [39 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Region of Enrollment [Number; unit: participants]
  France | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients in Non-progression at 2 Months
Description: Non-progression is defined as partial response, complete response or stable disease according to RECIST V1.0. Complete response is defined as the disappearance of all target lesions and partial response is defined as at least a 30% decrease in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline SLD (RECIST V1.0.).Stable disease is defined as no decrease or increase sufficient to qualify as partial response or progression with reference to SLD since the start of treatment. Radiologic assessment was carried out every 8 weeks.
Time Frame: 2 months
Population: 5 patients deceased at 2 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Efavirenz
Number analyzed (Participants) | 14
percentage of participants | 14.3 [1.8 to 42.8]

2. Secondary Outcome: Percentage of Patients in Non-progression at 4 Months
Description: as for outcome 1
Time Frame: 4 months
Population: 8 patients deceased at 4 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Efavirenz
Number analyzed (Participants) | 11
percentage of participants | 9.1 [0.2 to 41.3]

3. Secondary Outcome: Percentage of Patients in Non-biological Progression at 2 Months
Description: Non-biological progression was assessed using CA 19-9 every 28 days until end of treatment, and was defined as a 2-month CA19.9 concentration lower than 1.5 times the baseline CA 19-9 concentration.
Time Frame: 2 months
Population: 5 patients deceased at 2 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Efavirenz
Number analyzed (Participants) | 14
percentage of participants | 31.4 [4.7 to 50.8]

4. Secondary Outcome: Overall Survival
Description: OS was was defined as the time from the inclusion to death due to any cause. Participants without documented death were censored at the date of the last follow-up or last patient contact. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Through Database Cutoff Date of 06-July-2011 ( median follow-up time of 397 days)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efavirenz
Number analyzed (Participants) | 19
days | 216 [59 to 390]

5. Secondary Outcome: Event-free Survival
Description: Event-free survival (EFS) was defined as the delay between trial inclusion and the first of the following events: progression (biological or morphological), death, treatment interruption due to toxicity, initiation of another treatment. Morphological progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Biological progression is defined as a confirmed increase in CA 19-9 concentration to more than 1.5 times the baseline value, sustained over two consecutive monthly assessments.
  Patients without any of the aforementioned events at the time of the statistical analysis will be censored at the time they were last known to be event-free. The EFS was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Through Database Cutoff Date of 06-July-2011 ( median follow-up time of 397 days)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efavirenz
Number analyzed (Participants) | 19
days | 52 [22 to 56]

6. Secondary Outcome: Progression-free Survival
Description: Progression was defined as morphological or biological progression. Progression-free survival was defined as the delay between trial inclusion and progression (morphological or biological) or death for any reason. Morphological progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Biological progression is defined as a confirmed increase in CA 19-9 concentration to more than 1.5 times the baseline value, sustained over two consecutive monthly assessments. Patients who have not progressed nor died at the time of the statistical analysis will be censored at the time they were last known to be progression-free. The EFS was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Through Database Cutoff Date of 06-July-2011 ( median follow-up time of 397 days)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efavirenz
Number analyzed (Participants) | 19
days | 54 [23 to 56]

7. Secondary Outcome: Quality of Life Score
Description: EORTC-QLQ-C30 is a cancer-specific instrument with 30 questions to evaluate quality of life. The first 28 use a 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much) assessing 5 functional scales (physical, role, emotional, cognitive, social), 3 symptom scales (fatigue, nausea/vomiting, pain), six single symptoms (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties), and two global health/QoL questions. Items 29 and 30 use a 7-point scale (1=very poor to 7=excellent).Scores are linearly transformed from 0 to 100 per EORTC guidelines. Higher scores mean better functioning or QoL for functional/global scales, but worse symptoms for symptom scales and items. Score ranges (0-100): higher Functional scores = better QoL; higher Symptom scores= worse QoL; Higher Global health score= better QoL.
Time Frame: 2 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Efavirenz
Number analyzed (Participants) | 19
score on a scale
  Physical functionning score | 73.3 [53.3 to 100]
  Role functionning score | 75 [50 to 100]
  Emotional Functioning score | 83.3 [66.7 to 83.3]
  Cognitive Functioning score | 75 [66.7 to 100]
  Social Functioning score | 75 [50 to 100]
  Global health status score | 58.3 [50 to 83.3]
  Fatigue score | 44.4 [22.2 to 100]
  Nausea / Vomiting score | 0 [0 to 16.7]
  Pain score | 41.7 [0 to 66.7]
  Dyspnoea score | 33.3 [0 to 33.3]
  Insomnia score | 33.3 [0 to 66.7]
  Appetite loss score | 16.7 [0 to 66.7]
  Constipation score | 0 [0 to 66.7]
  Diarhoea score | 16.7 [0 to 66.7]
  Financial Problems score | 0 [0 to 33.3]

ADVERSE EVENTS:
Description: Only serious adverse events were monitored. Adverse events (non-serious) were not assessed/monitored during the study.
Arm/Group | Efavirenz
Serious Adverse Events (participants affected / at risk) | 12/19
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efavirenz (N=19)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Disease progression (General disorders) | 2 (2)
Pericardial constriction (Cardiac disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Euphoria (Psychiatric disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Biliary stent blockage (Hepatobiliary disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes